CLINICAL TRIAL: NCT02042170
Title: A Phase II, Multi-center, Randomized, Comparative, Parallel, Open, Dose Finding Study to Assess the Efficacy and Safety After 26 Week-treatment of Eutropin Plus (SR-hGH) Compared to Eutropin Inj. in Pre-pubertal Children With Idiopathic Short Stature
Brief Title: Efficacy and Safety Study of Sr-hGH in Comparison With Daily hGH in ISS Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: LG Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LG-SHCL010
Record Dates: First submitted 2014-01-20; First posted 2014-01-22 (Estimated); Last update posted 2016-03-24 (Estimated); Status verified 2015-09

CONDITIONS: Establishing Dose of Sr-hGH in ISS Patients

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Sr-hGH 0.5 mg/kg/wk (Experimental): Patients inject Eutropin plus (Sr-hGH) 0.5 mg/kg/wk every week himself/herself.
  Interventions: Drug: human growth hormone self-injection
- Sr-hGH 0.7 mg/kg/wk (Experimental): Patients inject Eutropin plus (Sr-hGH) 0.7 mg/kg/wk every week himself/herself.
  Interventions: Drug: human growth hormone self-injection
- Daily hGH 0.37 mg/kg/wk (Active Comparator): Patients inject Eutropin (daily hGH) 0.37 mg/kg/wk everyday for the first 6days a week himself/herself.
  Interventions: Drug: human growth hormone self-injection

INTERVENTIONS:
Drug: human growth hormone self-injection

SUMMARY:
The purpose of this study is to assess dosing requirements and establish the efficacy of SR-hGH in idiopathic short stature patients (ISS). This phase II study is designed as multi-center, randomized, active comparator-controlled, parallel, open-label.

45 patients were randomized to three arms with 1:1:1 ratio, two arms of Sr-hGH and one of daily hGH. Two doses of Sr-hGH were administered, which are 0.5 and 0.7mg/kg/week. And the other arm received daily hGH at 0.37 mg/kg/week.

Patients in Sr-hGH groups injected on a specific day of the every week for 26 weeks. And patients randomized to daily hGH group injected for 6 days a week.

Patients visited study centers five times, firstly at screening (Visit 1), at randomization (Visit 2), after 13th dosing (Visit 3), after 26th dosing (Visit 4), and finally for follow-up (Visit5).

ELIGIBILITY:
Criteria

* are older than or equal to age of 4
* are pre-pubertal (Tanner's stage I)
* are younger than bone age of 9 in female; of 11 in male
* have less than 3 years of a difference in bone and chronological age
* have confirmed idiopathic short stature

Ages: 4 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 46 (Actual)
Dates: Start 2014-02; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline in height velocity at Week 26, cm/year | Week 0-26

SECONDARY OUTCOMES:
Change from baseline in height velocity, cm/year | at Week 13
Change from baseline in height, cm | at Week 13 and 26
Change from baseline in IGF (Insulin-like growth factor)-I and IGF-I SDS (standard deviation score) | at Week 13 and 26

CONTACTS AND LOCATIONS:
Locations (1):
- Ho Sung Kim, Seoul, Seoul, South Korea